CLINICAL TRIAL: NCT03419910
Title: An Open-Label, Single-Sequence Study to Investigate the Effects of Cyclosporine on the Pharmacokinetics of BMS-986165 at Steady State in Healthy Male Participants
Brief Title: An Investigational Study of Cyclosporine on Experimental Medication BMS-986165 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-045
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986165 and cyclosporine (Experimental): BMS-986165 and cyclosporine administered orally
  Interventions: Drug: BMS-986165; Drug: Cyclosporine

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
Drug: Cyclosporine — Specified dose on specified days

SUMMARY:
This is an investigational study of Cyclosporine on the experimental medication BMS-986165 in healthy male participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participant, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body mass index 18.0 to 32.0 kg/m2
* Weight ≥ 50 kg

Exclusion Criteria:

* Any medical condition that presents a potential risk to the subject and/or may compromise the objectives of the study, including a history of or active liver disease
* History or presence of acute or chronic bacterial, fungal, or viral infection (eg, pneumonia, septicemia) within the 3 months prior to screening
* Known or suspected autoimmune disorder, or any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status
* History of administration of live vaccines within 60 days before screening
* Any history or risk for tuberculosis (TB)

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | 24 hours
Area under the concentration vs time curve from time zero to 24 hours post dose (AUC[0-24]) | 24 hours

SECONDARY OUTCOMES:
Adverse events (AEs) | Up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx